CLINICAL TRIAL: NCT04795453
Title: Assessment of Score System to Predict the Need for Surgery in Newborn Infants With Two and More Grades of NEC
Brief Title: Assessment of Score System of Surgery in Necrotizing Enterocolitis(NEC) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, director, Children's Hospital of Chongqing Medical University
Other Study IDs: NEC surgery
Record Dates: First submitted 2021-03-05; First posted 2021-03-12 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Necrotizing Enterocolitis; Neonate; Surgery
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- assessment of usual method to predict the need for surgery: two and more grades of NEC is assessed using the usual method to predict the need for surgery
  Interventions: Other: score system to predict the need for surgery; Other: usual method to predict the need for surgery
- assessment of score system to predict the need for surgery: two and more grades of NEC is assessed using the score system to predict the need for surgery
  Interventions: Other: score system to predict the need for surgery; Other: usual method to predict the need for surgery

INTERVENTIONS:
Other: score system to predict the need for surgery — two and more grades of NEC is assessed using the score system to predict the need for surgery
Other: usual method to predict the need for surgery — two and more grades of NEC is assessed using the usual method to predict the need for surgery

SUMMARY:
Necrotizing enterocolitis(NEC) is one of the most serious disease in the newborn infants, and two and more grades of NEC usually lead to surgery, even death. But, it is difficult to predict when to operate the surgery.

DETAILED DESCRIPTION:
Necrotizing enterocolitis(NEC) is characterized by vomit, abdominal distention, hypoactive bowel sounds and bloody stools, even shock, disseminated intravascular coagulation(DIC) and sepsis. X-ray is shown Intestinal wall gas and/or portal vein pneumatosis and pneumoperitoneum.

Two and more grades of NEC in newborn infant is a urgent condition, and whether or not operation is difficult to predict.

Here, the investigators develop a score system including five parameters(abdominal circumference, base excess, heart rate, severities of respiratory distress, sepsis) in one retrospective cohort, and the score system is used and assessed to predict the need for surgery in another prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* two and more of NEC is diagnosed in the newborn infants
* on the time of diagnosis for NEC both the surgery and non-surgery are reasonable according the surgeon's suggestions

Exclusion Criteria:

* pneumoperitoneum
* refusing to take part in the study according to parents' decision

Ages: 1 Hour to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: two and more of NEC is diagnosed in newborn infants during hospitalization
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
sensitivity of the score system for predicting the need of surgery | before surgery
  sensitivity of the score system for predicting the need of surgery is assessed
specificity of the score system for predicting the need of surgery | before surgery
  specificity of the score system for predicting the need of surgery is assessed
accuracy of the score system for predicting the need of surgery | before surgery
  accuracy of the score system for predicting the need of surgery is assessed
positive likelihood ratio of the score system for predicting the need of surgery | before surgery
  positive likelihood ratio of the score system for predicting the need of surgery is assessed
negative likelihood ratio of the score system for predicting the need of surgery | before surgery
  negative likelihood ratio of the score system for predicting the need of surgery is assessed
positive predictive value of the score system for predicting the need of surgery | before surgery
  positive predictive value of the score system for predicting the need of surgery is assessed
negative predictive value of the score system for predicting the need of surgery | before surgery
  negative predictive value of the score system for predicting the need of surgery is assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Chen（陈）, Chongqing, Chongqing Municipality, China